CLINICAL TRIAL: NCT04001985
Title: Nasogastric Tube Clamping Trial: Is it Useful? A Proposed Algorithm for Removal.
Brief Title: Nasogastric Tube Clamping Trial vs. Immediate Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Illinois College of Medicine at Peoria (Other)
Collaborators: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Robin Alley, Robin Alley MD, FACS Assistant Professor of Clinical Surgery, Assistant Program Director, University of Illinois College of Medicine at Peoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1429090-1
Record Dates: First submitted 2019-06-19; First posted 2019-06-28 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Small Bowel Obstruction; Ileus
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate NG tube removal (Active Comparator): Once the NG tube output is less than 500 mL over a 24 hour period with at least two other signs of return of bowel function the NG tube will be removed. Other signs of bowel function include flatus, bowel movement, change of NG tube output from bilious to more clear/frothy character, and hunger.
  Interventions: Other: No clamp trial
- NG tube clamp trial (Active Comparator): Once the NG tube output is less than 500 mL over a 24 hour period with at least two other signs of return of bowel function, a 4 hour clamp trial will be performed. Other signs of bowel function include flatus, bowel movement, change of NG tube output from bilious to more clear/frothy character, and hunger. The NG tube will be taken off of suction and clamped. The NG tube is then reconnected to suction at the end of the four hour clamp trial and removed if less 125 mL drains or kept in place if greater than 125 mL drains. The same initial criteria are used again to determine if a clamp trial will be performed after 24 hours.
  Interventions: Other: Clamp trial

INTERVENTIONS:
Other: No clamp trial — Once the NG tube output is less than 500 mL over a 24 hour period with at least two other signs of return of bowel function the NG tube will be removed. Other signs of bowel function include flatus, bowel movement, change of NG tube output from bilious to more clear/frothy character, and hunger.
  Arms: Immediate NG tube removal
Other: Clamp trial — Once the NG tube output is less than 500 mL over a 24 hour period with at least two other signs of return of bowel function, a 4 hour clamp trial will be performed. Other signs of bowel function include flatus, bowel movement, change of NG tube output from bilious to more clear/frothy character, and hunger. The NG tube will be taken off of suction and clamped. The NG tube is then reconnected to suction at the end of the four hour clamp trial and removed if less 125 mL drains or kept in place if greater than 125 mL drains. The same initial criteria are used again to determine if a clamp trial will be performed after 24 hours.
  Arms: NG tube clamp trial

SUMMARY:
The primary objective is to assess the need of clamping nasogastric tubes (NG) before removal. Outcomes of patients admitted requiring nasogastric tube decompression will be compared. Patients with small bowel obstruction (SBO), post-operative ileus, and ileus on admission that require nasogastric tube placement will be included in the study. The patients will be divided into two groups when return of bowel function is suspected based on set criteria for automatic removal of nasogastric tube versus nasogastric tube clamp trial.

Specific outcomes will be occurrence of nasogastric tube replacement, number of emeses if any, failure of clamp trial, aspiration pneumonia, and any other unplanned outcome.

DETAILED DESCRIPTION:
A high volume of patients are admitted to hospitals yearly for bowel obstruction/ileus complications. Lifetime risk of small bowel obstruction varies from 0.1%-5% if patients have not undergone abdominal surgery, but increases to 30% if the patient underwent a prior abdominal surgery. Ileus is also a common complication in the short term post-operative period. Both of these conditions are initially treated with nasogastric tube decompression if the patient is having emesis.

The investigators were unable to find any literature that shows a concrete volume of nasogastric tube output that was deemed the maximum for safe removal. Signs of return of bowel function can indicate it is safe to remove the nasogastric tube. These include flatus, bowel movements, decrease in nasogastric tube output amount, change of nasogastric tube output color from bilious (green) to more gastric (yellow) or salivary (clear/foamy) quality. Some physicians prefer to perform a clamp trial before removal of the nasogastric tube. The duration of the trial and cutoff amount of residual drainage varies among physicians. Regardless of the duration, the nasogastric tube is essentially stenting open the lower esophageal sphincter while it is left in place and not connected to suction. This, theoretically, places the patient at risk for aspiration and subsequent pneumonia. Information in the literature appears divided in regard to aspiration risk.

This study hopefully will support the statement that it is safe to remove the nasogastric tube with signs of bowel function, without the need for clamp trials and thus avoiding any possible adverse outcomes associated with the trial. The investigators also anticipate that this study will provide objective guidelines on which patients will continue to improve after nasogastric tube removal.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years or older
* Admitted under any of the teaching surgical services for small bowel obstruction or ileus, or develops post-operative ileus
* Patient agreeable to participation in the study

Exclusion Criteria:

* Under the age of 18
* Patient self-removes the NG requiring replacement will be removed from study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Necessity of replacement of NG tube | Through study completion, an average of 1 year
  This measure looks at if the NG tube is replaced in either arm of the study after removal.

SECONDARY OUTCOMES:
Pulmonary complications | Through study completion, an average of 1 year
  This outcome looks at any episodes of aspiration pneumonia, pneumonitis, or pneumothorax.
Days until discharge | Through study completion, an average of 1 year
  This outcome will look at the number of days until discharge for all patients in each arm.
Emesis episodes after NG tube removal | Through study completion, an average of 1 year
  This outcome is measured as the number of patients who had an episode of emesis after NG tube removal prior to discharge.
Days until general diet reached | Through study completion, an average of 1 year
  This outcome is measured by looking at how many days it takes from the time of ileus or SBO diagnosis to reach a general diet.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Alley, MD, Principal Investigator — University of Illinois College of Medicine at Peoria
Locations (1):
- OSF Saint Francis Medical Center, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhimanagouda V. G., Eshwar B. K., Hanumaraddi L. G., Mohammedgouse A. K. Early removal versus conventional removal of nasogastric tube after abdominal surgery: a prospective randomized controlled study. International Surgery Journal 4(1):220-232, 2017.
- [Background] Mamun K, Lim J. Role of nasogastric tube in preventing aspiration pneumonia in patients with dysphagia. Singapore Med J. 2005 Nov;46(11):627-31. PMID 16228094
- [Background] Mitchell CK, Smoger SH, Pfeifer MP, Vogel RL, Pandit MK, Donnelly PJ, Garrison RN, Rothschild MA. Multivariate analysis of factors associated with postoperative pulmonary complications following general elective surgery. Arch Surg. 1998 Feb;133(2):194-8. doi: 10.1001/archsurg.133.2.194. PMID 9484734
- [Background] Ibanez J, Penafiel A, Raurich JM, Marse P, Jorda R, Mata F. Gastroesophageal reflux in intubated patients receiving enteral nutrition: effect of supine and semirecumbent positions. JPEN J Parenter Enteral Nutr. 1992 Sep-Oct;16(5):419-22. doi: 10.1177/0148607192016005419. PMID 1433774
- [Background] McAlister FA, Bertsch K, Man J, Bradley J, Jacka M. Incidence of and risk factors for pulmonary complications after nonthoracic surgery. Am J Respir Crit Care Med. 2005 Mar 1;171(5):514-7. doi: 10.1164/rccm.200408-1069OC. Epub 2004 Nov 24. PMID 15563632
- [Background] Ferrer M, Bauer TT, Torres A, Hernandez C, Piera C. Effect of nasogastric tube size on gastroesophageal reflux and microaspiration in intubated patients. Ann Intern Med. 1999 Jun 15;130(12):991-4. doi: 10.7326/0003-4819-130-12-199906150-00007. PMID 10383370
- [Background] Izu BS, Monson B, Little AG, Termuhlen PM. Surgical practice: evidence or anecdote. J Surg Educ. 2009 Sep-Oct;66(5):281-4. doi: 10.1016/j.jsurg.2009.07.010. PMID 20005501
- [Background] Gero D, Gie O, Hubner M, Demartines N, Hahnloser D. Postoperative ileus: in search of an international consensus on definition, diagnosis, and treatment. Langenbecks Arch Surg. 2017 Feb;402(1):149-158. doi: 10.1007/s00423-016-1485-1. Epub 2016 Aug 3. PMID 27488952
- [Background] Fonseca AL, Schuster KM, Maung AA, Kaplan LJ, Davis KA. Routine nasogastric decompression in small bowel obstruction: is it really necessary? Am Surg. 2013 Apr;79(4):422-8. PMID 23574854
- [Background] Gomes CA Jr, Lustosa SA, Matos D, Andriolo RB, Waisberg DR, Waisberg J. Percutaneous endoscopic gastrostomy versus nasogastric tube feeding for adults with swallowing disturbances. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD008096. doi: 10.1002/14651858.CD008096.pub3. PMID 22419328
- See also: Epidemiology — https://online.epocrates.com/diseases/99323/Small-bowel-obstruction/Epidemiology